CLINICAL TRIAL: NCT01356732
Title: Determination of the 90% Effective Dose of a Sufentanil Bolus in Analgesia During Lateral Decubitus of Mechanically Ventilated Patients.
Acronym: REANURSUF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09 162 02
Record Dates: First submitted 2011-04-19; First posted 2011-05-19 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Pain
Keywords: mechanical ventilation; Midazolam; Ramsay; Sufentanil
MeSH Terms: conditions — Pain | interventions — Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sufentanil (Experimental)
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Sufentanil — From 0 to 0,05 µg/kg to a maximum of 4 µg/kg of sufentanil. 7 minutes before nursing 3 nursing per day during 3 days

SUMMARY:
Mechanically ventilated patients experiencing pain are frequent in intensive care units (ICU) however their treatment remains unclear. This prospective pharmacodynamic study relates to the analgesia of procedural pains. The primary objective was to determine the 90% effective dose (ED) of a sufentanil bolus to obtain a satisfactory analgesia (defined by a Behavioral Pain Scale (BPS) at 3 or 4) during lateral decubitus (LD) of mechanically ventilated patients.

Material and Method. Patients who, at rest before the 48th hour of mechanical ventilation, reach the objectives of BPS at 3 or 4 and Ramsay sedation score between 3 and 5, were included.

During a 72h evaluation phase, BPS was used to measure the efficiency of a bolus of sufentanil on the analgesia of the LD. The dose of this bolus was raised gradually every new LD until BPS was at 3 or 4.

ELIGIBILITY:
Inclusion Criteria:

* 48th hour of mechanical ventilation
* mechanical invasive ventilation
* 48th hour midazolam sedation
* Behavioral Pain Scale (BPS) at 3 or 4
* mechanical ventilation of 5 days duration

Exclusion Criteria:

* Pregnant or breast-feeding woman
* Impossibility of evaluation of the BPS tetraplegia, curare-link , post anoxic coma encephalic death
* Indication of deep conscious-sedation, malignant cranial trauma, toxic shock, acute respiratory distress syndrome
* Extra renal clearance OU people in hemodialysis
* Severe renal failure (creatinine clearance <15ml/min)
* Severe hepatic failure
* State of consciousness with impossibility to use self-assessment scale
* Body mass index >35 ou <18
* Sufentanil midazolam paracetamol allergy or contraindication
* Guardianship or confirmed criminal Subject who give his informed consent
* Morphinic other than sufentanil (morphine, alfentanil fentanyl, remifentanil, nalbuphine, codeine, buprenorphine)
* Antalgic other than sufentanil and paracetamol ( tramadol nefopam, ketamine, dextropropoxyphene, non steroidal anti-inflammatory drug )
* MAO inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The effective dose (ED) of a sufentanil bolus to obtain a satisfactory analgesia (defined by a Behavioral Pain Scale (BPS) at 3 or 4) | five days

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Fourcade, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Service de réanimation - Hôpital Purpan, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chaveron D, Silva S, Sanchez-Verlaan P, Conil JM, Sommet A, Geeraerts T, Genestal M, Minville V, Fourcade O. The 90% effective dose of a sufentanil bolus for the management of painful positioning in intubated patients in the ICU. Eur J Anaesthesiol. 2012 Jun;29(6):280-5. doi: 10.1097/EJA.0b013e328352234d. PMID 22388706